CLINICAL TRIAL: NCT04465942
Title: Immunotherapy in Lung Cancer: Which Treatment After Immunotherapy Cessation: A Prospective Registry From the European Lung Cancer Working Party
Brief Title: Immunotherapy in Lung Cancer: Treatment After IO Cessation.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: European Lung Cancer Working Party (Other)
Responsible Party: Sponsor
Other Study IDs: 01171
Record Dates: First submitted 2020-06-25; First posted 2020-07-10 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; Carboplatin; Pemetrexed; Paclitaxel; pembrolizumab; Nivolumab; atezolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: (chemo)immunotherapy — Patients are receiving immunotherapy or chemoimmunotherapy as a standard of care
  Other Names: cisplatinum; carboplatinum; pemetrexed; paclitaxel; pembrolizumab; nivolumab; atezolizumab

SUMMARY:
Immunotherapy is now a standard of care for first-line and eventually salvage therapy in patients with stage IV NSCLC and as adjuvant after RT-CT for stage III NSCLC.

The aim of the study is determining the therapeutic landscape and the reason for immunotherapy cessation.

DETAILED DESCRIPTION:
Patients with stage IV or unresectable not irradiable stage III NSCLC will be registered at the time receiving immunotherapy alone or in combination with chemotherapy.

When IO is stopped, reason for cessation and further treatment will be recorded.

Secondary endpoints are survival after IO cessation, activity of first salvage therapy, disease-free survival after IO cessation in patients receiving no further treatment.

Patients will be centrally registered at the ELCWP headquarter (Institut Jules Bordet, Brussels, Belgium).

ELIGIBILITY:
Inclusion Criteria:

* Histological diagnosis of non-small cell lung cancer (NSCLC)
* Stage IVA/IVB and unresectable and non irradiable stage III NSCLC naïve of immunotherapy.
* Patients who receive immunotherapy (any type) monotherapy, combined immunotherapy or in combination with chemotherapy for first or second-line treatment.
* Availability for participating in the detailed follow-up of the protocol.
* Signed informed consent.

Exclusion Criteria:

* Patients receiving adjuvant immunotherapy for stage I-III NSCLC are not eligible
* Tumours for which TNM stage at time of study inclusion cannot be assessed.
* History of prior malignant tumour, except non-melanoma skin cancer or in situ carcinoma of the cervix or of the bladder or cured malignant tumor (more than 5-year disease free interval).
* Any type of immunotherapy for previous cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IV or unresectable and non irradiable NSCLC, naïve of immunotherapy and receiving immunotherapy alone or combined chemo-immunotherapy
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-06-26 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
to determine the therapeutic landscape after cessation of an immune checkpoint therapy | From IO cessation date up to first treatment whatever the time in-between and up to 5 years
  Which treatment is proposed after IO cessation

SECONDARY OUTCOMES:
survival | From IO cessation date up to death or up to 5 years
  survival after ICI cessation, overall and in pre-defined subgroups (cessation for progressive disease [group 1], for toxicity [group 2], by patient decision without progression [group 3])
Activity of salvage therapy - response | At the end of cycle 2 or 3 (according to routine local practice), one cycle corresponding to 21 days, up to 6 cycles. assessment will done according to RECIST criteria
  Best response to first salvage chemotherapy after ICI
Disease-free survival | From IO cessation to progression documentation or death or up to 5 years
  disease-free survival in untreated non-progressive patients after ICI cessation
second-line ICI effectiveness - response | From initiation of second-line IO up to 2 years
  Response to second-line ICI (response rate) using WHO criteria
second-line ICI effectiveness - progression-free survival | From initation of second-line ICI up to progression or death and up to 5 years
  PFS to second-line ICI
Activity of salvage therapy - progression-free survival | From initation of salvage therapy up to progression or death and up to 5 years
  Progression-free survival to first salvage chemotherapy after ICI
Activity of salvage therapy - survival | From initation of second-line ICI up to death and up to 5 years
  Survival to first salvage chemotherapy after ICI

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Berghmans, MD, PhD, Study Chair — ELCWP
Locations (5):
- Belgium (5):
  - Department of Intensive Care Unit and Thoracic Oncology Institut Jules Bordet, Brussels
  - Department of Pneumology CHU Charleroi, Charleroi
  - Department of Pneumology Hôpital Saint-Joseph, Gilly
  - Hôpital Ambroise Paré, Mons
  - Hôpital Mont-Godinne, Yvoir

IPD SHARING:
Plan to Share IPD: Undecided